CLINICAL TRIAL: NCT03407170
Title: An Open-Label, Phase II Study to Determine the Immunologic Correlates of Pembrolizumab-Mediated Tumor Regression in Subjects With Advanced Melanoma (KEYNOTE-161)
Brief Title: Immunologic Determinants of Response to Pembrolizumab (MK-3475) in Advanced Melanoma (MK-3475-161/KEYNOTE-161)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-161; MK-3475-161 (Other: Merck); KEYNOTE-161 (Other: Merck)
Record Dates: First submitted 2018-01-18; First posted 2018-01-23 (Actual); Results first posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Advanced Melanoma
Keywords: Programmed Cell Death-1 (PD-1); PD1; Programmed Cell Death-Ligand 1 (PD-L1); Programmed Cell Death-Ligand 2 (PD-L2); PDL1; PDL2
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg by intravenous (IV) infusion every 3 weeks (Q3W) for up to 24 months
  Interventions: Biological: pembrolizumab

INTERVENTIONS:
Biological: pembrolizumab — 200 mg by IV infusion Q3W for up to 24 months
  Other Names: KEYTRUDA®; MK-3475

SUMMARY:
In this study, participants with advanced melanoma will be treated with pembrolizumab (MK-3475) and their tumors and blood will be analyzed for changes related to pembrolizumab therapy.

The primary hypotheses are that participants who respond to pembrolizumab have:

1. a higher fraction of cytotoxic tumor-infiltrating T-lymphocytes (FCT) at baseline compared to those who do not respond to pembrolizumab
2. a higher fold-increase in FCT compared to baseline than those who do not respond to pembrolizumab
3. a higher Average Specific Cytotoxic T-lymphocyte Frequency Ratio (ASCTFR) compared to those who do not respond to pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed diagnosis of unresectable stage III or metastatic melanoma not amenable to local therapy
* Has testing for a BRAF mutation prior to study entry
* Has measurable disease per RECIST 1.1 as assessed by the investigator/radiology
* Has resolution of toxic effect(s) of the most recent prior chemotherapy to Grade 1 or less (except alopecia). If the participant received major surgery or radiation therapy of >30 Gray units, they must have recovered from the toxicity and/or complications from the intervention
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 10 days of study start
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: is not a woman of childbearing potential (WOCBP) OR is a WOCBP and agrees to use a contraceptive method, consistent with local regulations regarding the methods of contraception for those participating in clinical studies, during the treatment period and for at least 120 days after the last dose of study treatment
* A male participant is eligible to participate if he agrees not to donate sperm PLUS to be abstinent from heterosexual intercourse as their preferred and usual lifestyle OR agree to use contraception, consistent with local regulations regarding the methods of contraception for those participating in clinical studies, during the treatment period and for at least 120 days after the last dose of study treatment

Exclusion Criteria:

* Has disease that is suitable for local therapy administered with curative intent
* Has a history of interstitial lung disease
* Has a positive pregnancy test within 72 hours before the first dose of study therapy
* Has received prior therapy with an anti-Programmed Cell Death Protein 1 (PD-1), anti-Programmed Cell Death-Ligand 1 (PD-L1), anti-Programmed Cell Death-Ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137)
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to study start
* Has received prior radiotherapy within 2 weeks of start of study therapy
* Has received a live vaccine within 30 days prior to the first dose of study therapy
* Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony stimulating factor [G-CSF], granulocyte macrophage colony stimulating factor [GMCSF] or recombinant erythropoietin) within 4 weeks prior to study start
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study therapy
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study therapy
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years with the exception of basal cell and squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study
* Is pregnant or breastfeeding or expecting to conceive or father children starting with the screening visit through 120 days after the last dose of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Massachusetts General Hospital ( Site 0102), Boston, Massachusetts
  - Dana Farber Cancer Institute ( Site 0101), Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg by intravenous (IV) infusion every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Zero participants are reported due to the risk of identification of a person.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg by IV infusion Q3W.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0
Age, Categorical [unit: Participants]
Sex: Female, Male [unit: Participants]
Ethnicity (NIH/OMB) [unit: Participants]
Race (NIH/OMB) [unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Mean Fraction of Cytotoxic T-lymphocytes (FCT) for Participants With Response Versus Participants With Progression
Description: FCT is defined as the fraction of CD8+ T-cells expressing a predefined single-cell ribonucleic acid (RNA) gene signature to the total tumor infiltrating CD8+T-cells isolated from tumor biopsies.
Time Frame: Up to approximately 59 weeks
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

2. Primary Outcome: Average Specific Cytotoxic T-lymphocyte Frequency Ratio (ASCTFR) for Participants With Response Versus Participants With Progression
Description: ASCTFR is defined as the arithmetic average of the log10 ratio of the frequency of individual specific cytotoxic T-Cell Receptor (TCR) clones of on-treatment to pre-treatment.
Time Frame: Up to approximately 59 weeks
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Baseline of Fraction of Cytotoxic T-lymphocytes (FCT) for Participants With Response Versus Participants With Progression
Description: The fold change from baseline in FCT. FCT is defined as the fraction of CD8+ T-cells expressing a predefined single-cell RNA gene signature to the total tumor infiltrating CD8+T-cells isolated from tumor biopsies.
Time Frame: Up to approximately 59 weeks
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 59 weeks
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Number of Participants Who Discontinued Any Study Drug Due to an Adverse Event (AE)
Description: The number of participants who discontinued any study treatment due to an AE is presented.
Time Frame: Up to approximately 59 weeks
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 1
Participants | 1

6. Secondary Outcome: Overall Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST Version 1.1 as assessed by the investigator.
Time Frame: Up to approximately 59 weeks
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS is defined as the time from start of treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurs first, per RECIST Version 1.1 as assessed by the investigator.
Time Frame: Up to approximately 59 weeks
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the start of treatment to death due to any cause.
Time Frame: Up to approximately 59 weeks
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Neoepitope Burden
Description: Neoepitope sequencing will be generated based on single cell ribonucleic acid (RNA) sequencing (scRNAseq), whole exome sequencing, and an epitope prediction algorithm to obtain neoepitope burden.
Time Frame: Up to approximately 59 weeks
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Antigenic Determinants of Highly-functional CD8 + T-cell Clones
Description: T-cell receptors (TCRs) from CD8+ T-cell clones will be identified by single cell ribonucleic acid (RNA) sequencing (scRNAseq) and their killing function will be confirmed by TCR-transduced T-cells recognizing autologous tumor-derived cell lines.
Time Frame: Up to approximately 59 weeks
Population: No data were collected or analyzed for this outcome measure due to early termination of the study.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 59 weeks
Description: Zero participants are reported due to the risk of identification of a person.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study was stopped early due to lack of accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT03407170/Prot_SAP_000.pdf